CLINICAL TRIAL: NCT02156843
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Safety and Efficacy of Pyridorin (Pyridoxamine Dihydrochloride) in Subjects With Nephropathy Due to Type 2 Diabetes (PIONEER)
Brief Title: Pyridorin in Diabetic Nephropathy
Acronym: PIONEER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: NephroGenex, Inc. (Industry)
Collaborators: Collaborative Study Group (CSG) (Network); Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PYR-311; 2014-001641-24 (EudraCT Number); CSG-17 (Other: Collaborative Study Group); PYR-311 (PIONEER) (Other: NephroGenex, Inc.)
Record Dates: First submitted 2014-05-28; First posted 2014-06-05 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Diabetic Nephropathy; Diabetic Kidney Disease
Keywords: Diabetic Kidney Disease; Nephropathy; Diabetic Nephropathy; Kidney Disease; Type 2 Diabetes
MeSH Terms: conditions — Diabetic Nephropathies; Kidney Diseases; Diabetes Mellitus, Type 2 | interventions — pyridoxamine dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pyridorin (Experimental): Pyridorin (pyridoxamine dihydrochloride) 300 mg oral BID (twice daily, every 12 hours) Capsule
  Interventions: Drug: Pyridorin
- Placebo (Placebo Comparator): Placebo Oral Capsule taken BID (twice daily, every 12 hours)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pyridorin — 300 mg BID (twice daily, every 12 hours), oral capsule taken until end stage renal disease or death occurs, or the study is terminated by the sponsor.
  Other Names: pyridoxamine dihydrochloride
  Arms: Pyridorin
Drug: Placebo — Placebo excipients without the active drug, oral capsule taken BID (twice daily, every 12 hours), until end stage renal disease or death occurs, or the study is terminated by the sponsor.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of oral Pyridorin 300 mg BID in reducing the rate of progression of nephropathy due to type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multi-center Phase 3 study to evaluate the safety and efficacy of Pyridorin 300 mg BID (twice daily, every 12 hours) in subjects with nephropathy due to type 2 diabetes mellitus. In this study, nephropathy is defined as a Serum Creatinine (SCr) >= 1.3 (≥1.25) mg/dL (111 umol/L) for female and >=1.5 (≥1.45) mg/dL (128 umol/L) for male subjects and a 24-hour urine collection protein/creatinine ration (PCR) >=1200 mg/g (136 mg/mmol), and if applicable for PS Phase, at Visit 1S or 1.1S a 24-urine collection PCR ≥600 mg/g (68 mg/mmol). Subjects must have a baseline SCr < 3.0 mg/dL (265 umol/L) and must be on previously established standard of care at screening.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting all of the following criteria will be eligible to participate in the study:

1. Patients who have given voluntary written informed consent to participate in this study prior to conducting Screening (Visit 1) procedures;
2. Patients 18 years of age or older with a diagnosis of type 2 diabetes;
3. Women of childbearing potential (WOCBP) who agree to use appropriate birth control (double-barrier methods, hormonal contraceptives, or intrauterine device) for the duration of the study (women of childbearing potential is defined as all women who are not surgically sterile or are not at least 1 year post menopausal). All women of childbearing potential must have a negative serum pregnancy test at Visit 1;
4. All men (unless surgically sterile, as defined below) who have sexual intercourse with a WOCBP must agree and commit to use a highly effective method of contraception for the duration of the study (defined as the time of the signing of the informed consent form through the conclusion of patient participation). Highly effective methods of contraception include:

   i. Male subjects agreeing that they and their female spouse/partners will use adequate contraception (2 forms of birth control, one of which must be barrier method) or be of non-childbearing potential.

   ii. To be considered surgically sterilized, a male partner must have had a vasectomy at least 24 weeks before Visit 1;
5. At Visit 1, patients must have a history of overt diabetic nephropathy, as defined by the following:

   * A SCr measurement ≥1.3 (≥1.25)mg/dL (111 µmol/L) for females or ≥1.5 (≥1.45) mg/dL (128 µmol/L) for males;
   * At Visit 1 or 1.1 24-hour urine collection PCR >1200 mg/g (130 mg/µmol) and, if applicable for PS phase, at Visit 1S or 1.1S a 24-urine collection PCR >600 mg/g (67 mg/µmol)
   * For eligibility determination, laboratory reported values of PCR will be rounded up to 2 significant digits (e.g. ≥1150 mg/g to 1200 mg/g; ≥595 mg/g to 600 mg/g),
6. Patients must have a SCr measurement <3.0 mg/dL (265 µmol/L);
7. Patients must have an eGFR of ≥20 mL/min/1.73m2, using the 4-variable Modification of Diet in Renal Disease equation in which eGFR = 175 x (SCr(mg/dL))-1.154 x (Age(years))-0.203 x (0.742 if female) x (1.212 if African American);
8. Patient must have a second screening SCr measurement at Visit 1.1 or 1.1S taken 1 week (± 2 days) after screening (Visit 1 or 1S). The value of the second screening SCr measurement must be <3.0 mg/dL (265 µmol/L) for both genders and within 25% of the first screening measurement;
9. Patients must be taking a single ACE-I or ARB at a constant dose for at least 26 weeks prior to Visit 1, where the dose of the ACE-I or the ARB is considered appropriate for that patient (can be zero to max dose approved by the FDA) and it is anticipated that the same dose can and will be maintained throughout the course of the study;
10. Patients taking any blood pressure medications in addition to an ACE-I or ARB, including diuretics, must be on a stable dose for 13 weeks prior to Visit 1 (and Visit 1S if applicable) with a seated blood pressure of ≤ 150/90 mmHg;
11. Patients not taking any blood pressure medications, including diuretics, other than an ACE-I or ARB must have a seated blood pressure ≤ 150/90 mmHg at Visit 1 (and Visit 1S if applicable) and a seated blood pressure considered appropriate for the patient and one that can be sustained throughout the study.

Exclusion Criteria:

Patients are excluded from participation in the study if any of the following criteria apply

1. Patients with type 1 diabetes or MODY (a monogenic form of diabetes);
2. Patients with a diagnosis of chronic kidney disease other than diabetic renal disease with or without hypertensive renal disease
3. Patients receiving a renin inhibitor or an aldosterone antagonist or a combination of an ACE-I and an ARB within 26 weeks of Visit 1
4. Patients with a history of solid organ transplantation
5. Patients with a history of myocardial infarction, coronary re-vascularization procedures (including percutaneous transluminal coronary angioplasty), stroke, or transient ischemic attack within 30 days prior to Visit 1
6. Patients with a diagnosis of New York Heart Association Class III or IV congestive heart failure at any time
7. Patients with a history of being treated for neoplastic disease (except basal or squamous cell carcinoma of the skin) within 5 years prior to Visit 1
8. Patients with any history of dialysis within 2 years prior to Visit 1
9. Patients in whom dialysis or renal transplantation is anticipated by their physician within 1 year after Visit 1
10. Patients who used SCr-altering drugs within 30 days prior to Visit 1
11. Patients who require systemic immunosuppression therapy for >2 weeks (except for inhalant steroids)
12. Patients with clinically significant liver disease or transaminase (alanine aminotransferase and aspartate aminotransferase) levels >2.5 × the upper limit of normal (ULN) measured at Visit 1.1 or Visit 1.1S
13. Patients with bilirubin levels >1.5 × ULN measured at Visit 1.1 or Visit 1.1S
14. Patients with a history of allergic or other adverse response to vitamin B preparations
15. Patients who require >50 mg of vitamin B6 daily
16. Patients who have an active history of dysphagia or swallowing disorders
17. Patients with a history of hypersensitivity to Pyridorin or any of the excipients (non-active ingredients) in the Pyridorin formulation
18. Patients who have taken pyridoxamine or any other investigational drug within 30 days prior to Visit 1, or have participated in a previous Pyridorin study or another interventional clinical study within 30 days prior to Visit 1
19. Patients with an active history of drug or alcohol abuse
20. Patients unlikely to comply with the study protocol (eg, an inability and unwillingness to participate in adequate training, an uncooperative attitude, inability to return for follow-up visits, or unlikelihood of completing the study)
21. Women who are lactating, pregnant, or intend to become pregnant during the course of the study
22. Persons employed with the sponsor, CRO, or one of the study investigative sites must be excluded from participation, even if they are not involved directly in the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2014-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Time to composite endpoint of >=50% SCr increase from baseline or ESRD | Approximately 45 Months
  Time to the composite endpoint consisting of the earliest event amongst a SCr increase of 50% from baseline that occurs during follow-up; or End Stage Renal Disease. ESRD is defined as the initiation of permanent dialysis, receiving a kidney transplant, or a SCr value >= 6.0 mg/dL (530 umol/L) with a second SCr confirmation value >=6.0 mg/dL (530 umol/L) obtained 4-6 weeks later. A confirmation of SCr value for subjects with ESRD and initiation of permanent dialysis or kidney transplant will not be collected.

SECONDARY OUTCOMES:
Time to the composite endpoint >=100% SCr increase or ESRD | Approximately 45 Months
  A SCr increase of >=100% that occurs during follow-up; or ESRD

OTHER OUTCOMES:
Change in serum cystatin-C | Change from baseline to Week 52 and from baseline to Week 104
Change in urine protein/creatinine ratio (PCR) | From baseline to Week 52 and from baseline to Week 104
Change in urinary transforming growth factor-beta (TGF-Beta) excretion | From baseline to Week 52 and from baseline to Week 104
Change in SCr | From baseline to Week 52 and from baseline to Week 104

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Dwyer, MD, Study Chair — The Collaborative Study Group (CSG) [Co-Chair]; Julia B. Lewis, MD, Study Chair — The Collaborative Study Group (CSG)
Locations (137):
- United States (55):
  - CSG Investigational Site (#157), Birmingham, Alabama
  - CSG Investigational Site (#130), Phoenix, Arizona
  - CSG Investigational Site (#150), Phoenix, Arizona
  - CSG Investigational Site (#145), Prescott, Arizona
  - CSG Investigational Site (#142), Tucson, Arizona
  - CSG Investigational Site (#160), Los Angeles, California
  - CSG Investigational Site (#143), Riverside, California
  - CSG Investigational Site (#159), Roseville, California
  - CSG Investigational Site (#153), Arvada, Colorado
  - CSG Investigational Site (#118), Aurora, Colorado
  - CSG Investigational Site (#120), Westminster, Colorado
  - CSG Investigational Site (#158), Waterbury, Connecticut
  - CSG Investigational Site (#156), Columbus, Georgia
  - CSG Investigational Site (#113), Chicago, Illinois
  - CSG Investigational Site (#102), Michigan City, Indiana
  - CSG Investigational Site (#115), New Orleans, Louisiana
  - CSG Investigational Site (#147), Greenbelt, Maryland
  - CSG Investigational Site (#117), Boston, Massachusetts
  - CSG Investigational Site (#114), Springfield, Massachusetts
  - CSG Investigational Site (#111), Detroit, Michigan
  - CSG Investigational Site (#134), Pontiac, Michigan
  - CSG Investigational Site (#162), Kansas City, Missouri
  - CSG Investigational Site (#152), Kansas City, Missouri
  - CSG Investigational Site (#141), Las Vegas, Nevada
  - CSG Investigational Site (#128), Buffalo, New York
  - CSG Investigational Site (#136), Northport, New York
  - CSG Investigational Site (#154), West Nyack, New York
  - CSG Investigational Site (#108), Asheville, North Carolina
  - CSG Investigational Site (#116), Charlotte, North Carolina
  - CSG Investigational Site (#125), Durham, North Carolina
  - CSG Investigational Site (#155), New Bern, North Carolina
  - CSG Investigational Site (#127), Winston-Salem, North Carolina
  - CSG Investigational Site (#124), Cincinnati, Ohio
  - CSG Investigational Site (#151), Cleveland, Ohio
  - CSG Investigational Site (#123), Cleveland, Ohio
  - CSG Investigational Site (#106), Columbus, Ohio
  - CSG Investigational Site (#148), Parma Heights, Ohio
  - CSG Investigational Site (#101), Philadelphia, Pennsylvania
  - CSG Investigational Site (#149), Pittsburgh, Pennsylvania
  - CSG Investigational Site (#146), Providence, Rhode Island
  - CSG Investigational Site (#131), Chattanooga, Tennessee
  - CSG Investigational Site (#105), Nashville, Tennessee
  - CSG Investigational Site (#119), Dallas, Texas
  - CSG Investigational Site (#139), Houston, Texas
  - CSG Investigational Site (#133), Houston, Texas
  - CSG Investigational Site (#109), Midland, Texas
  - CSG Investigational Site (#132), Salt Lake City, Utah
  - CSG Investigational Site (#107), Burlington, Vermont
  - CSG Investigational Site (#129), Charlottesville, Virginia
  - CSG Investigational Site (#137), Fairfax, Virginia
  - CSG Investigational Site (#103), Fairfax, Virginia
  - CSG Investigational Site (#104), Hampton, Virginia
  - CSG Investigational Site (#144), Richmond, Virginia
  - CSG Investigational Site (#121), Spokane, Washington
  - CSG Investigational Site (#122), Milwaukee, Wisconsin
- Australia (9):
  - CSG Investigational Site (#205), Camperdown, New South Wales
  - CSG Investigational Site (#201), Gosford, New South Wales
  - CSG Investigational Site (#206), Liverpool, New South Wales
  - CSG Investigational Site (#208), St Leonards, New South Wales
  - CSG Investigative Site (#204), Adelaide, South Australia
  - CSG Investigational Site (#207), Footscray, Victoria
  - CSG Investigational Site (#200), Reservoir, Victoria
  - CSG Investigational Site (#202), Richmond, Victoria
  - CSG Investigational Site (#209), Parkville
- Bulgaria (8):
  - CSG Investigational Site (#757), Plovdiv
  - CSG Investigational Site (# 750), Sofia
  - CSG Investigational Site (# 755), Sofia
  - CSG Investigational Site (# 756), Sofia
  - CSG Investigational Site (#751), Sofia
  - CSG Investigational Site (#752), Sofia
  - CSG Investigational Site (#753), Sofia
  - CSG Investigational Site (#754), Stara Zagora
- France (7):
  - CSG Investigational Site (#801), Grenoble, Cedex
  - CSG Investigational Site (#802), Paris, Cedex
  - CSG Investigational Site (#800), Boulogne-sur-Mer
  - CSG Investigational Site (#803), Colmar
  - CSG Investigational Site (#806), Montpellier
  - CSG Investigational Site (#804), Rhone
  - CSG Investigational Site (#805), Valenciennes
- Germany (8):
  - CSG Investigational Site (#709), Aschaffenburg
  - CSG Investigative Site (#702), Berlin
  - CSG Investigational Site (#706), Elsterwerda
  - CSG Investigational Site (#703), Heidelberg
  - CSG Investigational Site (#707), Herzberg
  - CSG Investigational Site (#701), Hoyerswerda
  - CSG Investigational Site (#708), Mainz
  - CSG Investigational Site (#700), München
- Hong Kong (3):
  - CSG Investigational Site (#400), Hong Kong
  - CSG Investigational Site (#402), Kwai Chung
  - CSG Investigational Site (#401), Shatin
- Hungary (13):
  - CSG Investigational Site (#501), Balatonfüred
  - CSG Investigational Site (#509), Budapest
  - CSG Investigational Site (#513), Budapest
  - CSG Investigational Site (#505), Budapest
  - CSG Investigational Site (#507), Debrecen
  - CSG Investigational Site (#508), Gyula
  - CSG Investigational Site (#502), Hatvan
  - CSG Investigational Site (#504), Kaposvár
  - CSG Investigational Site (#510), Kisvárda
  - CSG Investigational Site (#506), Pécs
  - CSG Investigational Site (#514), Székesfehérvár
  - CSG Investigational Site (#500), Szikszó
  - CSG Investigational Site (#503), Zalaegerszeg
- Israel (16):
  - CSG Investigational Site (#308), Safed, Zefad
  - CSG Investigational Site (#307), Ashkelon
  - CSG Investigational Site (#313), Beersheba
  - CSG Investigational Site (#300), Haifa
  - CSG Investigational Site (#304), Holon
  - CSG Investigational Site (#306), Jerusalem
  - CSG Investigational Site (#314), Jerusalem
  - CSG Investigational Site (#309), Kfar Saba
  - CSG Investigational Site (#302), Nahariya
  - CSG Investigational Site (#312), Petah Tikva
  - CSG Investigational Site (#315), Poria – Neve Oved
  - CSG Investigational Site (#311), Rishon LeZiyyon
  - CSG Investigational Site (#305), Tel Aviv
  - CSG Investigational Site (#303), Tel Aviv
  - CSG Investigational Site (#310), Tel Hasomer
  - CSG Investigational Site (#301), Ẕerifin
- CSG Investigational Site (# 850), Phoenix, Mauritius
- Poland (6):
  - CSG Investigational Site (#651), Bydgoszcz
  - CSG Investigational Site (#655), Chojnice
  - CSG Investigational Site (#653), Kielce
  - CSG Investigational Site (#657), Nowy Sącz
  - CSG Investigational Site (#652), Poznan
  - CSG Investigational Site (#656), Poznan
- Puerto Rico (3):
  - CSG Investigational Site (#112), Rio Piedras
  - CSG Investigational Site (#110), San Juan
  - CSG Investigational Site (#135), Toa Baja
- Spain (8):
  - CSG Investigational Site (#601), San Sebastián de los Reyes, Madrid
  - CSG Investigational Site (#605), Barcelona
  - CSG Investigational Site (#606), Barcelona
  - CSG Investigational Site (#603), Barcelona
  - CSG Investigational Site (#604), Barcelona
  - CSG Investigational Site (#600), Girona
  - CSG Investigational Site (# 607), Lleida
  - CSG Investigational Site (#602), Valencia